CLINICAL TRIAL: NCT04254718
Title: Preliminary Pilot Study of Digital Storytelling in the NICU
Brief Title: Digital Storytelling in the NICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Terrah Akard, Associate Professor, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 191469
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Bereavement
Keywords: NICU

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital Storytelling (Experimental): Legacy intervention via digital story for NICU parents
  Interventions: Behavioral: Digital Storytelling

INTERVENTIONS:
Behavioral: Digital Storytelling — Creation of a digital story about the infant with video and music selected by parents

SUMMARY:
Our long-term goal is to reduce suffering and long-term negative consequences for families in the Neonatal Intensive Care Unit (NICU). The overall purpose of this study is to test feasibility of a legacy intervention for NICU parents.

DETAILED DESCRIPTION:
Specific aims are:

(1) To determine the feasibility of a legacy intervention for NICU parents; and (2) to determine the feasibility of psychosocial instruments for NICU parents. We will recruit parents (N = 12) of 6 infants in the NICU who have received a palliative care consultation and expected to die by 1 year of age based on provider report. We will use a one-group pre- and post-test design. The intervention will be delivered by the PI or trained study staff conducting video-taped interviews with parents in private NICU rooms to create a digital story about their infant. The videographer will use the video and music selected by parents to create a digital story about the infant. The final digital story is provided to parents on a DVD or unlisted (private) YouTube link to keep. Parents will complete electronic psychosocial measures at enrollment (baseline/pre-intervention) and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Parents of infants in the NICU who have received a palliative care consult and expected to die by 1 year of age based on provider report:

  * Parent caregivers (ages 18 years and up) of infants
  * Parents will be defined as the legal guardians who act in the role of the infant's primary and secondary parent caregivers based on parent self-report.
* Able to speak and understand English
* Absence of cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in PROMIS Anxiety survey (short form) | Baseline and 1 month
  The PROMIS Anxiety (short form) survey measures the extent of anxiety. The range is 5-40, higher scores indicate higher anxiety
Change in PROMIS Depression Survey (short form) | Baseline and 1 month
  The PROMIS Depression survey measures the extent of depression. The range is 5-40, with 5 being least depressed and 40 being the most depressed.
Change in PROMIS Sleep Disturbance survey (short form) | Baseline and 1 month
  The PROMIS Sleep Disturbance instruments assess self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. Scores range from 4-20. Low scores indicate better sleep and high scores indicate worse sleep.
Change in PROMIS Meaning and Purpose survey (short form) | Baseline and 1 month
  The PROMIS Meaning and Purpose survey assess one's sense of life having purpose and that there are good reasons for living. Scores range from 6-30. Higher scores indicated perceptions of hopefulness, optimism, goal-directedness, and feelings that one's life is worthy.
Change in Benefit Finding Scale | Baseline and 1 month
  Benefit Finding Scale measures the degree of deriving positive growth from adversity. Scores range from 17-85 with high scores indicating more positive growth.

CONTACTS AND LOCATIONS:
Overall Officials: Terrah Akard, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nolensville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes